CLINICAL TRIAL: NCT00477789
Title: Effects of Allopurinol on Diastolic Function in Chronic Heart Failure Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universita di Verona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 802
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2007-05-24 (Estimated); Status verified 2007-05

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; diastolic dysfunction; uric acid
MeSH Terms: interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: allopurinol

SUMMARY:
In patients with chronic heart failure (CHF)due to dilated cardiomyopathy diastolic dysfunction occurs frequently and is related to a poor outcome. We have previously shown that parameters of diastolic function significantly correlate with uric acid levels, a marker of impaired oxidative metabolism. We aimed to determine whether inhibition of xanthine oxidase with allopurinol might affect diastolic function in patients with CHF.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure;
* left ventricular systolic dysfunction (ejection fraction <45%)
* stable clinical conditions in the previous three months
* optimal medical therapy for CHF
* normal sinus rhythm
* written informed consent
* age >18 years

Exclusion Criteria:

* renal failure (s-creatinine >2.5 mg/dl)
* already on allopurinol
* malignancies
* chronic inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
diastolic function uric acid levels BNP | three months

CONTACTS AND LOCATIONS:
Overall Officials: Mariantonietta Cicoira, MD, PhD, Principal Investigator — Division of Cardiology, University of Verona, Italy
Locations (1):
- Division of Cardiology, University Hospital of Verona, Verona, Italy